CLINICAL TRIAL: NCT00250003
Title: Preventive Home Visits for Healthy Pensioners- a Randomized Controlled Trial in Nordmaling
Brief Title: Preventive Home Visits for Healthy Pensioners- a Randomized Controlled Trial
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Umeå University (Other)
Collaborators: Ministry of Health and Social Affairs, Sweden (Other Government)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UmU2001:39
Record Dates: First submitted 2005-11-04; First posted 2005-11-07 (Estimated); Last update posted 2005-11-23 (Estimated); Status verified 2005-09

CONDITIONS: Prevention; House Calls
Keywords: Elderly; Preventive home visits

INTERVENTIONS:
Behavioral: Preventive home visits

SUMMARY:
To investigate whether preventive home visits for healthy persons 75+, made by professional health workers, can change the pattern of care utilization and if the quality of life can improve. The hypothesis is that care utilisation will reduce, mortality decrease and quality of life improve.

DETAILED DESCRIPTION:
To investigate whether preventive home visits for healthy pensioners aged 75 years and over , can change the pattern of care utilization and if the quality of life can improve. To investigate if the results will last after the intervention has come to an end.

The concept of care utilization can in this trial be clarified as:

* use of primary health care
* use of elderly care including elderly houses
* mortality
* use of hospital care

The concept of quality of life will in this trial be measured with a number of self judgements.

The trial is performed as a randomized controlled trial in a small rural community in the north of Sweden. The staff is professional health workers and the visits is performed in the pensioners own homes.

ELIGIBILITY:
Inclusion Criteria:

* older than 75 year
* living in their own home
* living in Nordmaling, Sweeden

Exclusion Criteria:

* any need of elderly care, long term care or frequent health care

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Dates: Start 2000-02; Study Completion 2001-12

PRIMARY OUTCOMES:
use of health care facilities during two years 2000-2001
all cause mortality during two years 2000 - 2001

SECONDARY OUTCOMES:
use of health care facilities 2002-2004
all cause mortality during 2002-2004

CONTACTS AND LOCATIONS:
Overall Officials: Lars Dahlgren, professor, Study Chair — Epeidemiology and Public Health, Umeå University
Locations (1):
- Umeå University, Epidemiology and Public Health, Umeå, Västerbotten County, Sweden